CLINICAL TRIAL: NCT02782091
Title: Validation of an Ecological Assessment of Executive Function (Multiple Errands Test) in Patients With Schizophrenia : Study of Discriminant Validity
Brief Title: Discriminant Validity of the Multiple Errands Test in Schizophrenia
Acronym: VALITEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P150701
Record Dates: First submitted 2016-05-17; First posted 2016-05-25 (Estimated); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Schizophrenia
Keywords: MET; Prognosis; Cognition; Ecological; Executive function
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Schizophrenia Patient (Experimental)
  Interventions: Behavioral: Multiple Errands Test (MET)
- Control Subject (Experimental)
  Interventions: Behavioral: Multiple Errands Test (MET)

INTERVENTIONS:
Behavioral: Multiple Errands Test (MET) — 1 hour assessment in an unknown district with 2 independent raters.
  Other Names: Errands Test (Shallice and Burgess, 1991)

SUMMARY:
Schizophrenia (SZ) is a chronic, severe disease resulting in a misperception of reality, major social withdrawal and cognitive disturbances. Executive dysfunctions are widely considered as primary determinants of functional outcome. However, classic neuropsychological executive function measures poorly represent patients' functional outcome and seem inappropriate to evaluate the real-world functional impact of the disease.

In this perspective, Shallice and Burgess have developed for brain-damaged patients, the Multiple Errands Test (MET) allowing to assess planning, adaptation, problem solving and mental flexibility in real life settings, thus better capturing day-to-day abilities and including contextual (social, perceptive) influences. Setting the assessment outside the laboratory can help to identify subtle executive impairment not systematically expressed in standard care conditions and consequently improve the future care solutions. MET is based on the Supervisory Attentional System model of executive functioning and attention control that specifies how thought and action schema become activated or suppressed for routine and non-routine circumstances.

MET has been designed to measure real-world executive performance confronting the participants to unpredictable affordances and interpersonal interactions while planning and problem solving. Patients are asked to accomplish several tasks of variable complexity in an unknown commercial district. Severals rules must be respected and thus an action plan, strategy formulation, time and space management with very little assistance of the examiner are required.

Most of the studies involving MET were conceived for patients with acquired brain damage. LeThiec offered an extensive protocol with the initial scoring system (in terms of inefficiencies, rule breaks, interpretation failures and task execution failures). Simplified versions of MET were also suggested to be more suitable in hospital settings. Only one study was done in SZ including a single patient, it is therefore difficult to draw conclusions about clinical utility in SZ. To date, no other studies investigated the suitability of MET in patients with psychosis, while executive impairment is well documented in this population The investigators hypothesized that the Multiple Errands Test (MET), an ecological assessment of executive function has a better ability to measure everyday adaptative functioning SZ, compared to conventional EF assessment methods.

DETAILED DESCRIPTION:
The objectives of this study are: (1) establish normative data and (2) study discriminant validity of this tool with a large panel of EF measures.

Methods:

60 clinically stable SZ patients and 60 controls will be administered MET, as well as two measures of executive function: Wisconsin Card Sorting Test - 64, 6 Elements Test. Functional outcome will be assessed through Behavioural Inventory of Executive Functioning (BRIEF-A), ECHELLES LAUSANNOISES D'AUTO-EVALUATION DES DIFFICULTES ET DES BESOINS (ELADEB scale) and Global Assessment of Functioning scale (GAF scale). Clinical measures will be recorded in patients (Positive And Negative Symptoms Scale (PANSS), State Trait Anxiety Inventory - Y (STAI-Y A), Diagnostic Interview for Genetic Studies (DIGS) and Family Interview for Genetic Studies (FIGS)).

Step1: The investigators will first compare patients and controls on all variables of MET and establish normative data.

Step 2: The investigators will then study the discriminant validity of MET. The investigators will compare MET with traditional measures of executive functioning. The investigators will assess the correlation between each executive measure and functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Experimental group
* Diagnosis of schizophrenia or schizoaffective disorder (DSM V criteria)
* Clinically stable
* Age : between18 and 50 years
* Social security affiliation
* French speakers
* Written consent signed

Control group

* Age : between18 and 50 years
* Social security affiliation
* French speakers
* Written consent signed

Exclusion Criteria:

* History of neurological or somatic disorders with sensori-motor impact
* Electroconvulsive therapy in the 6 months prior to participation
* Person living near the test site and/or knowing the neighborhood
* Person under guardianship
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Comparison of quantitative variable between score for MET and standard functional evaluation | Inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Franck SCHURHOFF, Prof, MD., Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No